CLINICAL TRIAL: NCT03730961
Title: A Randomized, Double-Blind, Placebo-Controlled, Cross-over Phase 2 Study of Continuous 8-Hour Intravenous Infusions of BMS-986231 in Patients With Heart Failure and Impaired Systolic Function Given a Standard Dose of Loop Diuretic
Brief Title: An Investigational Study of Continuous 8-Hour Intravenous Administrations of BMS-986231 in Participants With Heart Failure and Reduced Heart Function Given a Standard Dose of Loop Diuretic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV013-034; 2018-000970-31 (EudraCT Number)
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Results first posted 2021-01-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Failure; Myocardial Failure; Congestive Heart Failure; Heart Decompensation
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo+Diuretic to BMS-986231+Diuretic (Experimental): Administered in a cross over design with 8-hour continuous infusions and 7-28 day wash-out periods
  Interventions: Drug: BMS-986231; Drug: Furosemide; Drug: Placebo
- BMS-986231+Diuretic to Placebo+Diuretic (Experimental): Administered in a cross over design with 8-hour continuous infusions and 7-28 day wash-out periods
  Interventions: Drug: BMS-986231; Drug: Furosemide; Drug: Placebo

INTERVENTIONS:
Drug: BMS-986231 — Intravenous administration
Drug: Furosemide — Intravenous administration
Drug: Placebo — Intravenous administration

SUMMARY:
The purpose of this study is to investigate continuous 8-hour introductions of BMS-986231 in participants with heart failure and weakened heart function given a standard dose of diuretic.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Left ventricular ejection fraction <45%, as assessed by echocardiography, a multigated acquisition (MUGA) scan or magnetic resonance imaging (MRI) scan within 18 months
* On stable chronic guideline-directed therapy for HF including chronic loop diuretics, ACEi, ARBs, MRAs, ARNI or / and β-blockers as tolerated, with no changes of these medications in the past 2 weeks
* At least an oral dose of 40 mg of furosemide/day or equivalent (20 mg torsemide, 1 mg bumetamide)

Exclusion Criteria:

* SBP < 115 mm Hg or > 180 mm Hg at screening or pre-randomization
* Heart rate < 50 beats per minute (bpm) or > 120 bpm at screening or pre-randomization
* Primary HF etiology attributable to either restrictive/obstructive cardiomyopathy, idiopathic hypertrophic or uncorrected severe valvular disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United Kingdom (2):
  - Glasgow Clinical Research Facility, Glasgow
  - Richmond Pharmacology, London

REFERENCES:
- [Derived] Felker GM, Borentain M, Cleland JG, DeSouza MM, Kessler PD, O'Connor CM, Seiffert D, Teerlink JR, Voors AA, McMurray JJV. Rationale and design for the development of a novel nitroxyl donor in patients with acute heart failure. Eur J Heart Fail. 2019 Aug;21(8):1022-1031. doi: 10.1002/ejhf.1504. Epub 2019 Jun 6. PMID 31168885
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 participants were randomized/assigned to treatment, and 23 initiated period 1 treatment.
Groups:
- Sequence 1: First received placebo (period 1), then received BMS-986231 (period 2) following washout.
  Each treatment administered 8 hours continuous IV infusion at the dose of 12 μg/kg/min, corresponding to an infusion rate of 20 mL/H. At hour 4 after the start of the infusion, 40 mg IV bolus of furosemide administered through a separate IV line, given slowly over 1 to 2 minutes.
- Sequence 2: First received BMS-986231 (period 1), then received placebo (period 2) following washout.
  Each treatment administered 8 hours continuous IV infusion at the dose of 12 μg/kg/min, corresponding to an infusion rate of 20 mL/H. At hour 4 after the start of the infusion, 40 mg IV bolus of furosemide administered through a separate IV line, given slowly over 1 to 2 minutes.
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2
Started (Started = Initiated Period 1 treatment) | 12 | 11
Period 1 Completion | 12 | 11
Period 2 Completion | 11 (1 participant did not complete Period 2 due to hypotension but remained in the study) | 10 (1 participant discontinued study due to AE)
Completed (Completed study) | 12 | 10
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 8
  >=65 years | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.7 (8.19) | 69.8 (8.23) | 68.7 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 4-hour Urinary Output Following Intravenous Administration of 40 mg Furosemide to HFrEF Participants Receiving BMS-986231 Infusion Compared to Placebo
Description: The total volume of urinary output 4 hours after 40 mg furosemide bolus given to participants with HFrEF while on BMS-986231 compared to placebo: absolute difference in total volume and % change from placebo.
  Sequence 1: Placebo in period 1, drug in period 2
  Sequence 2: Drug in period 1, placebo in period 2
Time Frame: 4 hours
Population: Treated (per Protocol set) - All randomized participants who were given both study treatments and completed the study as per protocol. Participants are included in the treatment group they received in each period.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- BMS-986231: BMS-986231 administered 8 hours continuous IV infusion at the dose of 12 μg/kg/min, corresponding to an infusion rate of 20 mL/H. At hour 4 after the start of the infusion, 40 mg IV bolus of furosemide administered through a separate IV line, given slowly over 1 to 2 minutes.
- Placebo: Placebo administered 8 hours continuous IV infusion of D5W administered at the flow rate of 20 mL/H. At hour 4 after the start of the infusion, 40 mg IV bolus of furosemide administered through a separate IV line, given slowly over 1 to 2 minutes.
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 21 | 21
mL
  Sequence 1: number analyzed (Participants) | 11 | 11
  Sequence 1 | 900.7 (366.56) | 1603.3 (674.18)
  Sequence 2: number analyzed (Participants) | 10 | 10
  Sequence 2 | 1176.7 (386.21) | 1345.4 (391.11)
  Total | 1032.1 (392.74) | 1480.5 (559.92)
Statistical Analysis 1: Comparison: BMS-986231 vs Placebo; Test type: Superiority — Drug - placebo; p = 0.0021, t-test, 2 sided; Mean Difference (Net) = -448, 95% CI 2-sided [-714 to -183]
Statistical Analysis 2: Comparison: BMS-986231 vs Placebo; Test type: Superiority — Percent change Drug - placebo; p = 0.0222, t-test, 2 sided; Mean Difference (Net) = -22.1, 95% CI 2-sided [-40.7 to -3.51]

2. Secondary Outcome: FeNa in Participants With HFrEF While on BMS-986231 Compared to Placebo
Description: Secondary efficacy analyses was performed using the randomized population. The FeNa, FeK, furosemide urinary and plasma concentration and the ratio of urinary sodium to urinary furosemide was calculated at each time point over 4-hour urine/plasma collection after a bolus injection of 40 mg furosemide while receiving BMS-986231 or placebo.
  Fractional Excretion Na = ((Urine Sodium * Plasma Creatinine) / (Plasma Sodium * Urine Creatinine)) * 100
Time Frame: Day 1, predose; 0-4 hours, 4-5 hours, 5-6 hours, 6-7 hours, 7-8 hours
Population: All randomized subjects who started study drug infusion in at least one treatment period. This is also known as the Intent to Treat (ITT) population. Data in this data set was analyzed based on randomized sequence of treatments.
Measure: Mean (Standard Deviation); unit: percent of filtered sodium
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 23 | 23
percent of filtered sodium
  Before start of infusion: number analyzed (Participants) | 14 | 14
  Before start of infusion | 0.5 (0.52) | 0.6 (0.73)
  0-4 hours: number analyzed (Participants) | 15 | 16
  0-4 hours | 0.6 (0.67) | 0.7 (0.84)
  4-5 hours: number analyzed (Participants) | 17 | 17
  4-5 hours | 4.6 (3.34) | 5.4 (3.09)
  5-6 hours: number analyzed (Participants) | 18 | 14
  5-6 hours | 5.0 (2.87) | 7.0 (3.51)
  6-7 hours: number analyzed (Participants) | 16 | 18
  6-7 hours | 3.3 (2.33) | 4.7 (2.79)
  7-8 hours: number analyzed (Participants) | 18 | 15
  7-8 hours | 1.7 (1.26) | 3.3 (2.52)
Statistical Analysis 1: Comparison: BMS-986231 vs Placebo; Test type: Superiority — Drug - placebo, 0-4 hours after furosemide; p = 0.0163, t-test, 2 sided; Mean Difference (Net) = -4.25, 95% CI 2-sided [-7.63 to -0.876]
Statistical Analysis 2: Comparison: BMS-986231 vs Placebo; Test type: Superiority — Percent change Drug - placebo, 0-4 hours after furosemide; p = 0.2018, t-test, 2 sided; Mean Difference (Net) = -15, 95% CI 2-sided [-38.8 to 8.77]
Statistical Analysis 3: Comparison: BMS-986231 vs Placebo; Test type: Superiority — Drug - placebo, 0-8 hours after start of infusion; p = 0.0526, t-test, 2 sided; Mean Difference (Net) = -3.61, 95% CI 2-sided [-7.27 to 0.0446]
Statistical Analysis 4: Comparison: BMS-986231 vs Placebo; Test type: Superiority — Percent change Drug - placebo, 0-8 hours after start of infusion; p = 0.2076, t-test, 2 sided; Mean Difference (Net) = -14.9, 95% CI 2-sided [-38.8 to 9]

3. Secondary Outcome: FeK in Participants With HFrEF While on BMS-986231 Compared to Placebo
Description: Secondary efficacy analyses was performed using the randomized population. The FeNa, FeK, furosemide urinary and plasma concentration and the ratio of urinary sodium to urinary furosemide was calculated at each time point over 4-hour urine/plasma collection after a bolus injection of 40 mg furosemide while receiving BMS-986231 or placebo.
  Fractional Excretion K = ((Urine Potassium * Plasma Creatinine) / (Plasma Potassium * Urine Creatinine)) * 100
Time Frame: Day 1, predose; 0-4 hours, 4-5 hours, 5-6 hours, 6-7 hours, 7-8 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent of filtered potassium
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 23 | 23
percent of filtered potassium
  Before start of infusion: number analyzed (Participants) | 15 | 14
  Before start of infusion | 0.4 (0.16) | 0.4 (0.17)
  0-4 hours: number analyzed (Participants) | 16 | 16
  0-4 hours | 0.5 (0.20) | 0.4 (0.17)
  4-5 hours: number analyzed (Participants) | 17 | 17
  4-5 hours | 1.1 (0.67) | 0.9 (0.46)
  5-6 hours: number analyzed (Participants) | 18 | 14
  5-6 hours | 1.2 (0.54) | 1.2 (0.52)
  6-7 hours: number analyzed (Participants) | 16 | 18
  6-7 hours | 1.1 (0.42) | 1.0 (0.35)
  7-8 hours: number analyzed (Participants) | 18 | 15
  7-8 hours | 1.0 (0.32) | 0.8 (0.32)
Statistical Analysis 1: Comparison: BMS-986231 vs Placebo; Test type: Superiority — Drug - placebo, 0-4 hours after furosemide; p = 0.1621, t-test, 2 sided; Mean Difference (Net) = 0.431, 95% CI 2-sided [-0.189 to 1.05]
Statistical Analysis 2: Comparison: BMS-986231 vs Placebo; Test type: Superiority — Percent change Drug - placebo, 0-4 hours after furosemide; p = 0.0338, t-test, 2 sided; Mean Difference (Net) = 32, 95% CI 2-sided [2.72 to 61.3]
Statistical Analysis 3: Comparison: BMS-986231 vs Placebo; Test type: Superiority — Drug - placebo, 0-8 hours after start of infusion; p = 0.0600, t-test, 2 sided; Mean Difference (Net) = 0.766, 95% CI 2-sided [-0.0353 to 1.57]
Statistical Analysis 4: Comparison: BMS-986231 vs Placebo; Test type: Superiority — Percent change Drug - placebo, 0-8 hours after start of infusion; p = 0.0280, t-test, 2 sided; Mean Difference (Net) = 33.5, 95% CI 2-sided [4.02 to 63]

4. Secondary Outcome: Furosemide Urinary Concentrations
Description: Summary of urine recovery by interval, measured by amount excreted.
Time Frame: Day 1, predose, 0-2 hours, 2-4 hours, 4-5 hours, 5-6 hours, 6-7 hours, 7-8 hours, 8-10 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 23 | 23
mg
  Before start of infusion: number analyzed (Participants) | 11 | 10
  Before start of infusion | 0.2 (0.13) | 0.2 (0.11)
  0-2 hours: number analyzed (Participants) | 9 | 12
  0-2 hours | 0.1 (0.08) | 0.1 (0.11)
  2-4 hours: number analyzed (Participants) | 12 | 14
  2-4 hours | 0.3 (0.37) | 0.1 (0.11)
  4-5 hours: number analyzed (Participants) | 20 | 21
  4-5 hours | 7.9 (4.66) | 8.2 (4.56)
  5-6 hours: number analyzed (Participants) | 19 | 19
  5-6 hours | 4.3 (1.74) | 3.7 (1.48)
  6-7 hours: number analyzed (Participants) | 18 | 21
  6-7 hours | 2.8 (2.03) | 2.7 (1.43)
  7-8 hours: number analyzed (Participants) | 20 | 21
  7-8 hours | 2.0 (1.22) | 1.7 (1.15)
  8-10 hours: number analyzed (Participants) | 19 | 20
  8-10 hours | 1.7 (1.28) | 1.6 (1.00)

5. Secondary Outcome: Furosemide Plasma Concentrations
Description: Summary of plasma concentrations by interval.
Time Frame: Day 1: 4, 5, 6, 8, 10 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 23 | 23
ng/mL
  4 hours post-dose: number analyzed (Participants) | 12 | 11
  4 hours post-dose | 1605 (5384) | 63.6 (140.3)
  5 hours post-dose: number analyzed (Participants) | 21 | 20
  5 hours post-dose | 2049 (593.0) | 2145 (653.2)
  6 hours post-dose: number analyzed (Participants) | 21 | 21
  6 hours post-dose | 1122 (437.6) | 1146 (466.8)
  8 hours post-dose: number analyzed (Participants) | 21 | 21
  8 hours post-dose | 426.8 (204.8) | 476.6 (226.0)
  10 hours post-dose: number analyzed (Participants) | 22 | 19
  10 hours post-dose | 345.6 (386.6) | 244.3 (164.3)

6. Secondary Outcome: Ratio Urinary Sodium (Na) to Urinary Furosemide at 8 Hours Post-start Infusion
Description: Summary of urinary concentrations 0-4 hours after furosemide
  Ratio = Cumulative Sodium Excretion / Cumulative Furosemide in Urine
Time Frame: 0-4 hours after furosemide
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio of Urinary Na:Urinary furosemide
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 21 | 21
Ratio of Urinary Na:Urinary furosemide | 6.1 (3.18) | 10.1 (4.74)
Statistical Analysis 1: Comparison: BMS-986231 vs Placebo; Test type: Superiority; Difference between drug and placebo = -4.0, Standard Deviation 4.74

7. Secondary Outcome: Number of Participants With Clinically Relevant Hypotension
Description: Clinically relevant hypotension is defined as systolic blood pressure (SBP) < 90 mmHg or symptomatic hypotension during infusion
Time Frame: up to 8 hours
Population: Safety set : All randomized participants who take at least 1 dose of double-blind study treatment. Participants were included in the treatment group they received in each period.
Measure: Number; unit: Number of participants
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 23 | 23
Number of participants | 4 | 0

8. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: as for outcome 7
Time Frame: up to 8 days
Population: as for outcome 7
Measure: Number; unit: Number of participants
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 23 | 23
Number of participants | 8 | 6

9. Secondary Outcome: Number of Participants With an Abnormal Clinical Laboratory Value
Description: Number of participants who experienced an in-study abnormal clinical laboratory event under the category of Hematology, Chemistry or Urinalysis.
Time Frame: from first dose to 30 days post-last dose (ca. 5-8 weeks)
Population: as for outcome 7
Measure: Number; unit: Number of participants
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 23 | 23
Number of participants | 0 | 0

10. Secondary Outcome: Change From Baseline in Vital Signs - Blood Pressure
Description: The change in baseline for vital signs was reported for each arm.
Time Frame: Day 1, 8 hours post-dose (end of infusion)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 23 | 22
mmHg
  diastolic blood pressure | -14.5 (9.99) | -0.6 (10.46)
  systolic blood pressure | -28.4 (15.60) | -4.9 (14.55)

11. Secondary Outcome: Change From Baseline in Vital Signs - Heart Rate
Description: The change in baseline for vital signs was reported for each arm.
Time Frame: Day 1, 8 hours post-dose (end of infusion)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 22 | 22
beats/min | 0.5 (10.40) | -0.1 (8.08)

12. Secondary Outcome: Change From Baseline in Vital Signs - Oxygen Saturation
Description: The change in baseline for vital signs was reported for each arm.
Time Frame: Day 1, 8 hours post-dose (end of infusion)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: oxygen saturation percentage
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 23 | 22
oxygen saturation percentage | -1.0 (1.82) | 0.0 (1.56)

13. Secondary Outcome: Change From Baseline in Electrocardiograms (ECGs) - Mean Heart Rate
Description: The change in baseline for ECGs was reported for each arm.
Time Frame: Day 1, 8 hours post-dose (end of infusion)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 23 | 21
beats/min | 0.9 (7.97) | 1.6 (7.61)

14. Secondary Outcome: Change From Baseline in Electrocardiograms (ECGs) - PR, QRS Duration, QT, QTcF Intervals
Description: The change in baseline for ECGs was reported for each arm.
Time Frame: Day 1, 8 hours post-dose (end of infusion)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 23 | 21
msec
  PR Interval, Aggregate: number analyzed (Participants) | 15 | 15
  PR Interval, Aggregate | 2.0 (24.21) | -2.8 (12.17)
  QRS Duration, Aggregate | -0.9 (25.91) | 2.2 (21.46)
  QT Interval, Aggregate | -9.1 (27.88) | -7.9 (16.95)
  QTcF Interval, Aggregate | -11.2 (26.90) | -5.1 (16.74)

15. Secondary Outcome: Telemetry
Description: Telemetry data not collected.
Time Frame: Day 1, 8 hours post-dose
Population: Analysis population is 0, data not collected
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change From Baseline in Physical Examination - Body Weight
Description: The change in baseline for physical examinations was reported for each arm.
Time Frame: Day 1, 8 hours post-dose (end of infusion)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | BMS-986231 | Placebo
Number analyzed (Participants) | 20 | 19
kg | 0.2 (0.77) | -0.5 (0.72)

ADVERSE EVENTS:
Time Frame: From first dose to 100 days post-last dose (up to ca. 4 months)
Arm/Group | BMS-986231 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/23
Other Adverse Events (participants affected / at risk) | 6/23 | 3/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986231 (N=23) | Placebo (N=23)
Myocardial infarction (Cardiac disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986231 (N=23) | Placebo (N=23)
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 1
Hypotension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT03730961/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT03730961/SAP_001.pdf